CLINICAL TRIAL: NCT02097862
Title: An Open Label, Non-Randomized, Multi-Center Study To Assess The Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Intra-Discally in Patients With Degenerative Disc Disease
Brief Title: Adipose Cells for Degenerative Disc Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioheart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: ADI-US-DDD-001
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Degenerative Disc Disease
Keywords: Degenerative Disc Disease; Disc Disease; Back pain; stem cells; adipose stem cells; ADSCs
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Adipose Stem Cells — Injection of adipose derived stem cells intra-discally

SUMMARY:
The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe and 2) Is treatment effective in improving the disease pathology of patients with diagnosed degenerative disc disease.

DETAILED DESCRIPTION:
This will be an open-label, non-randomized, multi-center study of ASC implantation performed intra-discally. ASCs will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells.

The adipose tissue specimen will be collected from the patient's abdomen using a liposuction cannula. In addition, a sample of peripheral blood will be collected for isolation of platelet rich plasma. The adipose tissue is processed for separation of the adipose tissue-derived stem cells, which are then resuspended in platelet rich plasma and transferred for intra-discal administration. The number of cells injected will vary depending on the amount of tissue processed and the number of cells obtained from the process. Following the injections follow-up data will be collected 3, 6 and 12 months after treatment.

Total study time frame is anticipated to be approximately 6 months. This study will enroll approximately 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative disease of one, two, or three lumbar discs with predominant back pain after conservative treatment (physical and medical) for over 6 months.
* Fibrous ring capable of holding the cell implantation, demonstrated by RMI image
* Absence of spinal infection.
* Haematological and biochemical analysis with no significant alterations that contraindicates intervention.
* The patient is able to understand the nature of the study.
* Informed written consent of the patient.

Exclusion Criteria:

* Congenital or acquired diseases leading to spine deformations that may upset cell application.
* Spinal segmental instability, spinal canal stenosis, isthmus pathology and other conditions that may compromise the study
* Modic III changes on MRI images (31).
* More than 50% loss of height
* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. Patients known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis will have an expert consultation as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg or greater than 180mmHg
* Resting heart rate > 100 bpm;
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Active clinical infection
* Unwilling and/or not able to give written informed consent.
* Recent smoking history or substance abuse (within six weeks)
* Use of > 20 alcoholic drinks per week
* Patients on Plavix or equivalent platelet inhibitors

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 12 months
  This is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot be directly measured.

SECONDARY OUTCOMES:
Oswestry | 12 months
  Low back questionnaire designed to determine how low back pain has affected your daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- US Stem Cell Clinic, Sunrise, Florida, United States

REFERENCES:
- [Background] Comella K, Silbert R, Parlo M. Effects of the intradiscal implantation of stromal vascular fraction plus platelet rich plasma in patients with degenerative disc disease. J Transl Med. 2017 Jan 13;15(1):12. doi: 10.1186/s12967-016-1109-0. PMID 28086781